CLINICAL TRIAL: NCT04127383
Title: Effectiveness, Cost-effectiveness and Implementation of the Assessment of Burden of Chronic Conditions (ABCC)-Tool in Patients With COPD, Asthma, Diabetes Mellitus Type 2 and Heart Failure: a Pragmatic Clustered Quasi-experimental Study
Brief Title: Effectiveness and Implementation of the Assessment of Burden of Chronic Conditions (ABCC)-Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Netherlands Instititute for Health Services Research (Other); TNO (Other); University of Twente (Other)
Responsible Party: Principal Investigator, Esther Boudewijns, Principal investigator, Maastricht University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-10400-98-001
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Diabetes Mellitus, Type 2; Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Diabetes Mellitus, Type 2; Heart Failure

STUDY DESIGN:
Intervention Model Description: Pragmatic clustered quasi-experimental study
Who Masked: Outcomes Assessor
Masking Description: Blinding of healthcare providers and patients is not possible due to the nature of the intervention, but the study team will be blind to treatment arms in the data set during data cleaning, handling of missing data, statistical analyses and drawing of conclusions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABCC-tool (Experimental): The intervention group will use the ABCC-tool during consultation with their healthcare provider. Healthcare providers in the intervention group will receive a short instructional film about the ABCC-tool before the start of the study. Additionally, healthcare providers from 12 practices will be invited for interviews, evaluating the context and process of implementation.
  Interventions: Device: Assessment of Burden of Chronic Conditions (ABCC)-tool
- Usual care (No Intervention): The control group will receive usual care, and healthcare providers will not be instructed

INTERVENTIONS:
Device: Assessment of Burden of Chronic Conditions (ABCC)-tool — The tool consists of a questionnaire, a visualisation using balloons, and treatment advice. A patient completes the questionnaire before consultation. The questionnaire measures the experienced burden of the chronic condition(s), and several risk factors. The questionnaire consists of a generic part and disease-specific parts. The generic questionnaire will be combined with any amount of disease-specific questionnaires (i.e. COPD, asthma, diabetes type 2 and heart failure), to form a single personalised scale and balloon chart for each individual patient. Outcomes of the questionnaire are visualised using balloons. The healthcare provider opens the visualisation during consultation. A balloon represents a domain, and the colour and height indicate a score on that domain. If a patient and healthcare provider select a balloon by clicking on it, treatment advice is shown by means of pop-ups. Based on the discussion following treatment advice, personal care plans can be determined.
  Arms: ABCC-tool

SUMMARY:
This study is designed to evaluate the effectiveness and implementation of the Assessment of Burden of Chronic Conditions (ABCC)-tool for patients with COPD, asthma, diabetes mellitus type 2 or heart failure (and any combination of these conditions) in real-life routine practice. The ABCC-tool consists of a questionnaire, a visualisation using balloons that is based on cut-off points, and treatment advice. The ABCC-tool is intended to be used in daily healthcare practice, is designed to monitor a patient's integrated health status over time, to facilitate shared decision making, and to stimulate self-management. The study has a pragmatic clustered quasi-experimental design with two arms. The intervention group will use the ABCC-tool and the control group will receive usual care. The study will be implemented at a general practice-level, and has a follow-up period of 18 months. The primary outcome is change in perceived quality of care, as measured with the Patient Assessment of Chronic Illness Care (PACIC), as compared to usual care after 18 months. It is hypothesized that the change in perceived quality of care is significantly higher in the group using the ABCC-tool as compared to the group that receives usual care. Additionally the implementation of the ABCC-tool in general practices will be evaluated in 12 general practices. The implementation study will evaluate the context of caregivers with the Consolidated Framework for Implementation Research, the process of implementation with the RE-AIM framework, and fidelity to the intervention with the fidelity framework.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis COPD, asthma, Diabetes Mellitus type 2 and/or heart failure
* can understand and read the Dutch language

Exclusion Criteria:

* COPD or asthma: used prednisone due to an exacerbation less than six weeks ago
* Heart failure or diabetes mellitus type 2: hospitalized less than six weeks ago
* Healthcare providers or patients who have already used the Assessment of Burden of COPD-tool are excluded from the control group
* Patients who have already used the Assessment of Burden of COPD-tool will be excluded from the intervention group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Perceived quality of care (PACIC): Patient Assessment of Chronic Illness Care | 0 months (baseline), 18 months
  Measured with the Patient Assessment of Chronic Illness Care, for total group. The scale has 20 items. Answers range from 1 to 5. Average scores (range 1-5) will be calculated. Higher scores mean more frequent presence of the aspect of structured chronic care.

SECONDARY OUTCOMES:
Perceived quality of care (PACIC): Patient Assessment of Chronic Illness Care | 0 months (baseline), 6 months, 12 months
  Measured with the Patient Assessment of Chronic Illness Care, for total group and for each condition separately. The scale has 20 items. Answers range from 1 to 5. Average scores (range 1-5) will be calculated. Higher scores mean more frequent presence of the aspect of structured chronic care.
Perceived quality of care (PACIC): Patient Assessment of Chronic Illness Care | 0 months (baseline), 18 months
  Measured with the Patient Assessment of Chronic Illness Care, for each condition separately. The scale has 20 items. Answers range from 1 to 5. Average scores (range 1-5) will be calculated. Higher scores mean more frequent presence of the aspect of structured chronic care.
Quality of life (EQ-5D-5L) | 0 months (baseline), 6 months, 12 months, 18 months
  Measured with the EuroQol-5D-5L, for total group and for each condition separately. The scale consists of the EQ-5D-5L descriptive system with 5 questions, and a VAS-scale. Answers range from 1 (best) to 5 (worst). EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, will be converted into a single index value (Dutch values). The EQ-5D-5L VAS will also be determined.
Capability well-being (ICECAP-A) | 0 months (baseline), 6 months, 12 months, 18 months
  Measured with the ICEpop CAPability measure for Adults, for total group and for each condition separately. The questionnaire consists of 5 questions. Answers range from 1 (no capability) to 4 (full capability for an attribute). A tariff value for an overall state can be calculated by summing the values across the individual attributes. This code will allow calculation of ICECAP-A tariffs for each respondent in a study
Patients' activation (PAM) | 0 months (baseline), 6 months, 12 months, 18 months
  Measured with the Patient Activation Measure, for total group and for each condition separately. The questionnaire consists of 13 questions on a 5-point scale. The scores range from 0 to 100. The higher the score, the more capable a person is in self-management.
Medical Consumption within Health Care | 0 (baseline), 3, 6, 9, 12, 15 and 18 months
  Measured with the Medical Consumption Questionnaire (MCQ), for total group and for each condition separately. The questionnaire includes 16 questions related to frequently occurring contacts with health care providers. The items will be valued using standard cost prices in the Netherlands. The costs of medical consumption are calculated by multiplying the volumes of care by the cost per unit of care. This will be used for a cost-effectiveness analysis.
Productivity losses | 0 (baseline), 3, 6, 9, 12, 15 and 18 months
  Measured with the Productivity Costs Questionnaire (PCQ), for total group and for each condition separately. The questionnaire includes 9 questions related to the impact of disease on the ability of a person to perform work. The items will be valued using standard cost prices in the Netherlands. Productivity lossess are calculated by multiplying the volumes by cost prices per unit. This will be used for a cost-effectiveness analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Onno CP van Schayck, Prof., Study Director — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data can be shared with researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Peters LH, Joore MA, Gidding-Slok AH, Keijsers LC, Twellaar M, Boudewijns EA, van Schayck OC, Muris JW, Kimman ML. Cost-effectiveness analysis of the Assessment of Burden of Chronic Conditions (ABCC) tool in primary care in the Netherlands. BMJ Open. 2025 Jun 24;15(6):e099762. doi: 10.1136/bmjopen-2025-099762. PMID 40555443
- [Derived] Boudewijns EA, Claessens D, van Schayck OCP, Twellaar M, Winkens B, Joore MA, Keijsers LCEM, Krol S, Urlings M, Gidding-Slok AHM. Effectiveness of the Assessment of Burden of Chronic Conditions (ABCC)-tool in patients with asthma, COPD, type 2 diabetes mellitus, and heart failure: A pragmatic clustered quasi-experimental study in the Netherlands. Eur J Gen Pract. 2024 Dec;30(1):2343364. doi: 10.1080/13814788.2024.2343364. Epub 2024 May 13. PMID 38738695
- [Derived] Boudewijns EA, Claessens D, Joore M, Keijsers LCEM, van Schayck OCP, Winkens B, Gidding-Slok AHM. Effectiveness and cost-effectiveness of the Assessment of Burden of Chronic Conditions (ABCC) tool in patients with COPD, asthma, diabetes mellitus type 2 and heart failure: protocol for a pragmatic clustered quasi-experimental study. BMJ Open. 2020 Nov 17;10(11):e037693. doi: 10.1136/bmjopen-2020-037693. PMID 33203626
- See also: Related Info — https://software.memic.maastrichtuniversity.nl/ziektelastmeter/